CLINICAL TRIAL: NCT00226525
Title: Rate of Metal Skin Allergy in Cohorts of Patients With and Without Coronary Stent Restenosis
Brief Title: Effect of Metal Skin Sensitivity on Restenosis After Stent Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 20-03.09.04-HMO-CTIL
Record Dates: First submitted 2005-07-10; First posted 2005-09-27 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-09

CONDITIONS: Coronary Stent Restenosis
Keywords: Restenosis, skin metal allergy

INTERVENTIONS:
Procedure: skin sensitivity test

SUMMARY:
This trial is intended to find wether there is a connection between allergy to metals and reooclusion of stents in the coronary arteries

ELIGIBILITY:
Inclusion Criteria:

Patients with 2 cardiac catheterization in one years time and in the first one stent implantation

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-02; Study Completion 2006-08

PRIMARY OUTCOMES:
The rate of skin delayed type hypersensitivity to metals among patients with restenosis and without restenosis

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Durst, MD, Principal Investigator — Cardiology Department Hadassah Medical Center Jerusalem Israel
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel